CLINICAL TRIAL: NCT06047964
Title: A Prospective, Multicenter, Clinical Trial to Evaluate the Safety and Effectiveness of the Intracranial Paclitaxel Drug-eluting Balloon Catheters (SeQuent® Please CIS) in the Endovascular Treatment of Symptomatic Intracranial Atherosclerotic Stenosis and Restenosis After Interventional Therapy
Brief Title: SeQuent ® Please CIS for the Treatment of INtracranial Atherosclerotic Stenosis
Acronym: SPINAS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: B. Braun Medical International Trading Company Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SPINAS
Record Dates: First submitted 2023-08-30; First posted 2023-09-21 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-09

CONDITIONS: Stroke; Intracranial Atherosclerotic Stenosis
Keywords: symptomatic intracranial atherosclerotic stenosis; DCB
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- De-novo DCB group (Experimental): Patients with de-novo symptomatic intracranial atherosclerotic stenosis and treated with DCB
  Interventions: Device: DCB
- De-novo POBA group (Active Comparator): Patients with de-novo symptomatic intracranial atherosclerotic stenosis and treated with POBA
  Interventions: Device: POBA
- Restenosis group (Experimental): Patients with symptomatic intracranial atherosclerotic re-stenosis after interventional therapy and treated with DCB
  Interventions: Device: DCB

INTERVENTIONS:
Device: DCB — Intracranial paclitaxel drug-eluting balloon catheters (SeQuent® Please CIS)
  Arms: De-novo DCB group; Restenosis group
Device: POBA — Intracranial PTA balloon catheter
  Arms: De-novo POBA group

SUMMARY:
This study is aiming to evaluate the safety and efficacy of SeQuent® Please CIS in the endovascular treatment of symptomatic intracranial atherosclerotic stenosis and restenosis after interventional therapy.

DETAILED DESCRIPTION:
This study includes 2 sub-studies, sub-study A and sub-study B, namely.

Sub-study A is a prospective, multicenter, randomized controlled, superior clinical trial to evaluate the safety and effectiveness of paclitaxel drug-releasing intracranial balloon catheter (SeQuent® Please CIS) in the treatment of symptomatic intracranial atherosclerotic stenosis.

Sub-study B is a prospective, multicenter, single-arm clinical trial designed to evaluate the safety and efficacy of paclitaxel drug-releasing intracranial balloon catheter (SeQuent® Please CIS) for the treatment of restenosis following interventional treatment for symptomatic intracranial atherosclerotic stenosis.

A total of 277 subjects are expected to be enrolled, including 252 subjects in sub-study A and 25 subjects in sub-study B. Subjects enrolled in sub-study A will be randomized into the study arm and the control arm with the ratio of 1:1. The study arm will be treated with SeQuent® Please CIS (paclitaxel drug-releasing intracranial balloon catheter), while the control arm will be treated with intracranial PTA balloon catheter. Subjects enrolled in sub-study A will all be treated with SeQuent®, Please CIS.

All subjects will be followed up till 12 month post procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 to 80 years old (including boundary value), gender is not limited;
2. The target lesion of the patient is a symptomatic intracranial atherosclerotic stenosis lesion (for part A only) or restenosis lesions after interventional therapy (for part B only);
3. Symptomatic intracranial arterial stenosis (intracranial segment of internal carotid artery (Petrous segment and above), middle cerebral artery, intracranial segment of vertebral artery, basilar artery, etc.) within 6 months, the degree of stenosis of the diseased artery is between 70% and 99% (WASID method);
4. Patients with symptoms occurring more than once (symptoms refer to stroke or transient ischemic attacks) after intensive drug therapy of internal medicine (including antiplatelet therapy, antihypertensive therapy, hypoglycemic therapy and lipid-lowering therapy);
5. The intracranial arterial stenosis lesion to be treated is a single lesion;
6. Patients with at least 1 risk factor for intracranial atherosclerotic plaque, including previous or existing hypertension, hyperlipidemia, diabetes, smoking;
7. Preoperative mRS ≤ 2, and NIHSS≤8;
8. Patients whose life expectancy is greater than 12 months as assessed by the investigator.
9. Patients or their guardians can understand the trial purpose, voluntarily participate in and sign the informed consent form, and can accept follow-up visits.

Exclusion Criteria:

1. Severe calcification in the target vessel, severe distortion of the target vessel or anatomical factors that make it hard for interventional devices to be in place;
2. Ischemic symptoms are only associated with branch events;
3. Severe stenosis or occlusion of tandem extracranial or intracranial vessels at the proximal or distal end of the target vessel;
4. Angioplasty or stenting procedures is planned for extracranial vascular lesions with tandem intracranial vessels;
5. History of endarterectomy in the extracranial segment of carotid artery and vertebral artery within 30 days;
6. The target vessel has previously been treated with stenting or angioplasty or other mechanical devices (for Part A only);
7. Acute or subacute intraluminal thrombosis is found in the target vessel;
8. Patients with intracranial stenosis combined with aneurysm, intracranial tumor or intracranial vascular malformation, or intracranial arterial spasm without significant stenosis;
9. Intracranial hemorrhage (cerebral intraparenchymal hemorrhage, massive subarachnoid hemorrhage, and subdural/epidural hemorrhage) within 3 months;
10. There are cardiogenic stroke or risk factors that may contribute to cardioembolism, such as fibrillation, left ventricular thrombosis or myocardial infarction within 6 weeks,;
11. Patients with abnormal coagulation function or bleeding tendency (e.g., international normalized ratio (INR) > 1.5);
12. Patients with known hypersensitivity to iodine contrast medium, paclitaxel, or iopromide;
13. Patients who are participating in clinical trials of other drugs or devices;
14. Other conditions that the investigator deems the patient unsuitable for enrollment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 281 (Actual)
Dates: Start 2023-03-23 (Actual); Primary Completion 2024-09-29 (Actual); Study Completion 2025-01-23 (Estimated)

PRIMARY OUTCOMES:
restenosis incidence of target lesion | 6 months post-procedure
  angiographic restenosis measured by WASID ( Warfarin-Aspirin Symptomatic Intracranial Disease) method in core-lab

SECONDARY OUTCOMES:
Device success rate | baseline procedure
  Successful delivery, dilatation and withdraw of the balloon
The changes of Modified Rankin Scale(mRS) score | 6 and 12 months post-procedure
  Scores range from 0 to 6, with higher scores indicating more severe nerve damage; Change of mRS score = mRS score at 6 months (12 months) after surgery - mRS score at baseline
The changes of NIH Stroke Scale(NIHSS) score | 6 and 12 months post-procedure
  Scores range from 0 to 42, with higher scores indicating more severe nerve damage; Change of NIHSS score = NIHSS score at 6 months (12 months) after surgery - NIHSS score at baseline.
Number and incidence (%) of target vessel stroke events (including ischemic or hemorrhagic stroke), transient ischemic attack | 6 and 12 months post-procedure
  Incidence of target vessel stroke events (%) = (number of subjects with target vessel stroke events/total number of subjects) × 100%.
  Incidence of transient ischemic attacks (%) = (number of subjects with transient ischemic attacks/total number of subjects) × 100%.
Recurrence incidence of ipsilateral ischemic stroke | 30 days, 6 and 12 months post-procedure
  Recurrence incidence of ipsilateral ischemic stroke (%) = (number of subjects with recurrent ipsilateral ischemic stroke/total number of subjects) × 100%.

CONTACTS AND LOCATIONS:
Overall Officials: Liqun Jiao, MD, Principal Investigator — Xuanwu Hospital, Beijing; Yan Ma, MD, Principal Investigator — Xuanwu Hospital, Beijing
Locations (9):
- China (9):
  - Xuanwu Hospital, Capital Medical University, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - Nanyang Central Hospital, Nanyang, Henan
  - The First Hospital of Jilin University, Changchun, Jilin
  - Jining First People's Hospital, Jining, Shandong
  - The Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - Renji Hospital, Shanghai Jiaotong University, School of Medicine, Shanghai, Shanghai Municipality
  - First Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - The Second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No